CLINICAL TRIAL: NCT03681431
Title: Phase II Clinical Trial to Evaluate an Antibiotic Regimen Pharmacokinetic Applicable to Outpatient Parenteral Antimicrobial Therapy in Enterococcus Faecalis Infective Endocarditis
Brief Title: Evaluation of an Antibiotic Regimen Pharmacokinetic Applicable to Enterococcus Faecalis Infective Endocarditis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ENDOKINETIC-CEF
Record Dates: First submitted 2018-08-03; First posted 2018-09-24 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Infectious Endocarditis
Keywords: Pharmacokinetic; Ceftriaxone; Enterococcus faecalis; Infectious Endocarditis
MeSH Terms: conditions — Endocarditis, Subacute Bacterial | interventions — Ceftriaxone

STUDY DESIGN:
Intervention Model Description: A phase II, single-centre, open, non-randomized, cross-over, clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ceftriaxone 4g/ 24h (Experimental): Single intravenous dose of Ceftriaxone 4g/ 24h
  Interventions: Drug: Ceftriaxone 4g/ 24h
- Ceftriaxone 2g/ 12h (Active Comparator): Two intravenous doses of Ceftriaxone 2g/ 12h
  Interventions: Drug: Ceftriaxone 2g/ 12h

INTERVENTIONS:
Drug: Ceftriaxone 4g/ 24h — Each individual will be administrated 2 doses of 2 g of ceftriaxone separated for 12 hours. After a wash-out period (5-7 days) the same individuals will receive a single dose 4 g of ceftriaxone. In both cycles, plasma drug concentrations will be measure during 24 hours.
  Arms: Ceftriaxone 4g/ 24h
Drug: Ceftriaxone 2g/ 12h — Each individual will be administrated 2 doses of 2 g of ceftriaxone separated for 12 hours. After a wash-out period (5-7 days) the same individuals will receive a single dose 4 g of ceftriaxone. In both cycles, plasma drug concentrations will be measure during 24 hours.
  Arms: Ceftriaxone 2g/ 12h

SUMMARY:
The clinical trial is designed as a phase II, crossover clinical trial. It will be carried out in healthy volunteers, who will receive two different antibiotic regimen based on ceftriaxone. One of the regimens had shown clinical effectiveness in this scenario, but it is not suitable for OPAT programs. In the other hand, a new treatment schema useful in OPAT programs is proposed, but there is still a lack of pharmacokinetic data to support it. The plasma drug concentrations will be measured in both cases, comparing the minimal drug concentration observed and the pharmacokinetic profiles of the two regimens.

DETAILED DESCRIPTION:
Infective endocarditis (IE) is an uncommon but virulent infection disease. One of the most frequent etiology for this infection is Enterococcus faecalis. IE treatment is difficult due to the characteristics of the infection itself, the bacterial species and the frequent comorbidities of the patients. A bactericidal antimicrobial treatment is mandatory for the resolution of this disease, but most antibiotics do not exhibit this effect against E. faecalis and have prompted the combination of an aminoglycoside and a cell-wall active agent (generally a β-lactam) as the standard treatment. This is a lengthy treatment (4-6 weeks) and its primary side effect is nephrotoxicity. Furthermore, aminoglycoside resistant strain's rates are increasing in USA and Europe, getting more complicated to establish an effective antibiotic regimen. Nowadays, patients with E. faecalis IE are old and often have significant underlying comorbidities with an increased risk of developing nephrotoxicity with aminoglycoside treatment. For this reason, and for the relevance of high-level aminoglycoside-resistant strains, some alternatives have been explored. A double β-lactam regimen is an option, despite the intrinsically resistance of E. faecalis to cephalosporins. The most studied combination is a regimen based on ampicillin plus ceftriaxone, which has shown a synergistic effect in vitro. This combination is as effective as ampicillin plus gentamycin, but with lower nephrotoxicity. Those patients need at least 4-6 weeks of treatment with a prolonged hospitalization. However, after 2 week of treatment some patients are clinically stabilized and could be benefit of an outpatient parenteral antibiotic therapy (OPAT) program. For that purpose, it is essential to design a treatment regimen, which ensures the effectiveness and safety of the treatment, based on stability and pharmacokinetic and pharmacodynamics (PK/PD) studies of the administered drugs. Furthermore, the logistic and schedule should be simple enough to enable the inclusion in an OPAT program. In order to design an antibiotic regimen suitable for OPAT programs and as effective as the standard therapies for E. faecalis IE, we decided to start clinical trial.

The clinical trial is designed as a phase II, crossover clinical trial. It will be carried out in healthy volunteers, who will receive two different antibiotic regimen based on ceftriaxone. One of the regimens had shown clinical effectiveness in this scenario, but it is not suitable for OPAT programs. In the other hand, a new treatment schema useful in OPAT programs is proposed, but there is still a lack of pharmacokinetic data to support it. The plasma drug concentrations will be measured in both cases, comparing the minimal drug concentration observed and the pharmacokinetic profiles of the two regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults subjects.
2. Weight between 40 and 105 kilograms, both included, and body mass index lower than 34 kilograms per square meter.
3. The subject (or his/her "trusted representative") must have given his/her informed and signed consent approved by an Ethical Committee.
4. The subject must have normal analytical values or abnormal without clinical significance of biochemical parameters, liver and kidney function panel test, hemogram and album level. A medical check will be run by workers of Infectious Diseases Department.
5. The subject must have a normal physical examination or abnormal without clinical significance. A medical check will be run by workers of Infectious Diseases Department.
6. The medication taken usually by the subjects will be check by the Pharmacy Department in order to find possible interactions with ceftriaxone.

Exclusion Criteria:

1. Subjects with clinically significant abnormalities in laboratory test or physical exploration. A medical check will be run by workers of Infectious Diseases Department.
2. Subjects undergoing an active infection find at the screening.
3. Subjects with any clinical or surgery condition which contraindicate his/her inclusion, check by workers of Infectious Diseases Department.
4. Subjects who has received treatment with cephalosporins 21 days before the trial starts or during the trial (apart from the protocol treatment).
5. Subjects hypersensitive or allergic to cephalosporines or penicillins.
6. Subjects undergoing chronic or acute cutaneous diseases which prevent the treatment administration.
7. Subjects not giving his/her informed and signed consent approved by an Ethical Committee.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Serum levels after 24 hours | 24 hours
  To determinate whether 24 hours after the administration of 4 grams of ceftriaxone in a single short infusion, serums levels would be higher than 5 micrograms per millilitre

SECONDARY OUTCOMES:
AUC 24 hours | 24 hours
  To compare the 24 hours area under the curve (AUC) after the administration of 4 grams of ceftriaxone in a single short infusion and the administration of 2 grams of ceftriaxone in a two short infusions separated for 12 hours.
Plasma Clearance | 24 hours
  To determinate ceftriaxone plasma clearance after the administration of 4 grams of ceftriaxone in a single short infusion.
Elimination Half-life | 24 hours
  To determinate ceftriaxone elimination half-life after the administration of 4 grams of ceftriaxone in a single short infusion.
Volume of Distribution | 24 hours
  To determinate ceftriaxone volume of distribution after the administration of 4 grams of ceftriaxone in a single short infusion.
Maximum Plasma Concentration | 24 hours
  To determinate ceftriaxone maximum plasma concentration after the administration of 4 grams of ceftriaxone in a single short infusion.
Safety: Number, frequency and importance of adverse reactions. | 1 month
  To determinate the safety (number, frequency and importance of adverse reactions) of the administration of 4 grams of ceftriaxone in a single short infusion

CONTACTS AND LOCATIONS:
Overall Officials: Maria Victoria H Gil Navarro, Principal Investigator — University Hospital Virgen del Rocio/ Institute of Biomedicine of Seville
Locations (1):
- University Hospital Virgen del Rocio, Seville, Spain

DOCUMENTS (1):
  • Study Protocol (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT03681431/Prot_000.pdf